CLINICAL TRIAL: NCT03421886
Title: Assessment of the Efficacy of Orthodontic Tooth Movement Using the Aerodentis System
Brief Title: Assessment of the Efficacy of the Aerodentis System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Chung How Kau, Professor and Chair, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160418007
Record Dates: First submitted 2018-01-12; First posted 2018-02-05 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Orthodontic Treatment; Tooth Crowding; Orthodontics
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Aerodentis system (Experimental): 30 patients will be systematically assigned to the treatment group (wearing Aerodentis Device).
  Interventions: Device: Aerodentis system
- Invisalign clear aligner system (Active Comparator): 15 patients will be systematically assigned to the control group (wearing clear aligners).
  Interventions: Device: Invisalign clear aligner system

INTERVENTIONS:
Device: Aerodentis system — The Aerodentis system is intended for the treatment of tooth malocclusion and is treated by applying force, over time, to teeth requiring alignment. It is an individually-fitted, plastic dental mouthpiece that is inserted and worn by the patient according to the dental practitioner's treatment plan. The Aerodentis system is comprised of a plastic mouthpiece containing an inflatable balloon that provides pressure (force) on the selected teeth designated to be moved to a final treated state. The inflatable balloon is inflated to the desired pressure using an electrical air pump unit that is programmed by the dental practitioner using Dror Orthodesign proprietary software; thus creating a course treatment specially designed for each patient.
  Arms: Aerodentis system
Device: Invisalign clear aligner system — Clear aligners are used for the treatment of tooth malocclusion. In these devices, a series of mouthpieces are used, where the force created by each mouthpiece on the treated teeth is designed to push the teeth in small, one step increments, toward the desired result.
  Arms: Invisalign clear aligner system

SUMMARY:
The purpose of this study is to evaluate the efficacy of the Aerodentis System for orthodontic tooth movement in an open label, two-arms, non-inferiority clinical study. This open-label, two-arm study will follow 45 patients for up to fifteen months. Thirty participants will wear the Aerodentis device, and fifteen participants will wear Invisalign, a commonly used clear appliance. Patients will be assigned to participate in the treatment group using the Aerodentis device at home for 10 hours daily or in the control group using clear correctors for the duration of up to 15 months. Outcome assessments will be performed every 4 weeks. Assessments will include tooth movement and quality of life assessments.

DETAILED DESCRIPTION:
The Aerodentis system is intended for the treatment of tooth malocclusion and is treated by applying force, over time, to teeth requiring alignment. Traditionally, the force has been created by attaching brackets to the teeth and creating tension through the stretching of flexible wire connected between the brackets. Alternatively, aligners are used for the treatment of tooth malocclusion. In these devices, a series of mouthpieces are used, where the force created by each mouthpiece on the treated teeth is designed to push the teeth in small, one step increments, toward the desired result.The Aerodentis system is comprised of a plastic mouthpiece containing an inflatable balloon that provides pressure (force) on the selected teeth designated to be moved to a final treated state. The inflatable balloon is inflated to the desired pressure using an electrical air pump unit that is programmed by the dental practitioner using Dror Orthodesign proprietary software; thus creating a course treatment specially designed for each patient.

A participant is required to wear the Aerodentis device or conventional clear correctors. Initial photos of participants will be reviewed to establish a pool of eligible potential participants. Then participants will be randomly selected for one of the two groups. Those wearing the Aerodentis device will be asked to answer a quality of life questionnaire. Follow-up assessments will be conducted every 4 weeks for both Aerodentis participants and clear corrector participants. During these assessment's we will look at movement of teeth, any side effects or discomfort the individual may be facing, patient assessment of whether the Aerodentis device is used regularly. Both intraoral and extraoral photos will be taken of patients, during certain time points of the study, as requested by PI or sponsor. If a participant enters and completes the entire study, then that individual will be in the study for up to 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Permanent dentition
* Patients that in the opinion of the investigator will be compliant with device use. Compliance is determined by patient questionnaire.
* Class I malocclusion with crowding of <6 mm between the anterior teeth from the right first premolar to the left first premolar, on the upper and lower.
* Good oral hygiene, as determined by investigator orthodontist.

Exclusion Criteria:

* Any medical or dental condition that, in the opinion of the investigator, could negatively affect study results during the expected length of the study. Conditions can include poor oral hygiene, extensive dental treatments, or periodontal disease.
* Patient is currently using any investigational drug or any other investigational device.
* Patient plans to relocate or move during the treatment period.
* Pregnant females. Orthodontic treatment is not advised in pregnant females.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chung How Kau, BDS, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Wang J, Lamani E, Christou T, Li P, Kau CH. A randomized trial on the effects of root resorption after orthodontic treatment using pulsating force. BMC Oral Health. 2020 Aug 27;20(1):238. doi: 10.1186/s12903-020-01226-z. PMID 32854693

RESULTS

PARTICIPANT FLOW:
Groups:
- Aerodentis System: 30 patients was systematically assigned to the treatment group (wearing Aerodentis Device).
  Aerodentis system: The Aerodentis system is intended for the treatment of tooth malocclusion and is treated by applying force, over time, to teeth requiring alignment. It is an individually-fitted, plastic dental mouthpiece that is inserted and worn by the patient according to the dental practitioner's treatment plan. The Aerodentis system is comprised of a plastic mouthpiece containing an inflatable balloon that provides pressure (force) on the selected teeth designated to be moved to a final treated state. The inflatable balloon is inflated to the desired pressure using an electrical air pump unit that is programmed by the dental practitioner using Dror Orthodesign proprietary software; thus creating a course treatment specially designed for each patient.
- Invisalign Clear Aligner System: 15 patients was systematically assigned to the control group (wearing clear aligners).
  Invisalign clear aligner system: Clear aligners are used for the treatment of tooth malocclusion. In these devices, a series of mouthpieces are used, where the force created by each mouthpiece on the treated teeth is designed to push the teeth in small, one step increments, toward the desired result.
Period: Overall Study
Arm/Group | Aerodentis System | Invisalign Clear Aligner System
Started | 30 | 15
Completed | 23 | 13
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Aerodentis System: 28 patients was systematically assigned to the treatment group (wearing Aerodentis Device) due to 2 run-in fails.
  Aerodentis system: The Aerodentis system is intended for the treatment of tooth malocclusion and is treated by applying force, over time, to teeth requiring alignment. It is an individually-fitted, plastic dental mouthpiece that is inserted and worn by the patient according to the dental practitioner's treatment plan. The Aerodentis system is comprised of a plastic mouthpiece containing an inflatable balloon that provides pressure (force) on the selected teeth designated to be moved to a final treated state. The inflatable balloon is inflated to the desired pressure using an electrical air pump unit that is programmed by the dental practitioner using Dror Orthodesign proprietary software; thus creating a course treatment specially designed for each patient.
- Total: Total of all reporting groups
Arm/Group | Aerodentis System | Invisalign Clear Aligner System | Total
Number analyzed (Participants) | 30 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (12) | 32.3 (16.4) | 31 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 10 | 35
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Litter's Index (Change in Little's Index Mean Total Score From Baseline)
Description: The Litter's Index of Displacement score is the primary clinical endpoint used to judge patient success. Tooth alignment is assessed by Litter's Index of Displacement. It is performed at the five contact points for the teeth located in lower 1's through 3's. This index is the sum of the numbers recorded at each of the 5 points which are in millimeters.
  Subjects were followed for a total of up to 15 months or until achieving a Little's index of <1.5, whichever came first. The Litter's Index was performed at the baseline and the end-point of the study.
  Data was analyzed by comparing the Baseline Little's Index with statistical analysis between investigational and control groups, and the Final Little's Index between investigational and control groups. Comparison of change in Little's Index from baseline to final was also done between investigational and control groups.
  A negative change in from baseline to the end-point represent a decrease in the degree of anterior irregularity.
Time Frame: Movement was recorded by capturing the start and end point of the 6 anterior teeth before and at the completion of the treatment respectively. Changes was compared and assessed. The duration of the treatment was an average of 10 months.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Aerodentis System | Invisalign Clear Aligner System
Number analyzed (Participants) | 23 | 13
mm
  Baseline Little's Index | 5.7 (2.3) | 6.2 (2.9)
  Endpoint Little's Index | 0.6 (0.5) | 0.3 (0.3)
  Change of Little's Index | -3.9 (2.8) | -4.7 (2.8)

ADVERSE EVENTS:
Time Frame: 55 weeks (13.75 months)
Arm/Group | Aerodentis System | Invisalign Clear Aligner System
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/15
Other Adverse Events (participants affected / at risk) | 0/30 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT03421886/SAP_000.pdf
  • Study Protocol (2016-07-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT03421886/Prot_001.pdf
  • Informed Consent Form (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT03421886/ICF_002.pdf